CLINICAL TRIAL: NCT02467998
Title: The Registry of Negative Pressure Wound Therapy for Chronic Wounds and Ulcers
Brief Title: Negative Pressure Wound Therapy Registry
Acronym: NPWTR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: U.S. Wound Registry (Other)
Responsible Party: Sponsor
Other Study IDs: CDR003
Record Dates: First submitted 2014-11-24; First posted 2015-06-10 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Foot Ulcers; Venous Stasis Ulcer; Pressure Ulcer; Surgical Wound Dehiscence; Burns; Other Types of Chronic Non Healing Wounds
Keywords: meaningful use; electronic health records; structured language; NPWT; PQRS
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Surgical Wound Dehiscence; Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NPWT treated wounds: NPWT from any FDA cleared NPWT device including
  Interventions: Device: NPWT

INTERVENTIONS:
Device: NPWT — SVAP polyurethane foam, RENASYS foam, RENASYS gauze, AMD gauze, VAC white sponge, VAC black sponge, applied with various NPWT devices, in addition to various dressings to protect wound edges
  Other Names: the VAC; Renasys; Pico; Engenix; Sved; SNaP; extriCARE; Prospera; Invia Liberty; Invia Motion; Avance; Halo MINI; COBALTT; Halo XT

SUMMARY:
The goal of the Negative Pressure Wound Therapy Registry (NPWTR) for Wounds is to provide real world patient data from electronic health records submitted to meet Stage 2 Meaningful Use in order to understand the effectiveness and safety of various NPWT devices and methods among patients with chronic wounds and ulcers. Randomized, controlled trials to establish product efficacy routinely exclude patients with the co-morbid conditions common to patients seen in usual clinical practice and thus the results of these Randomized Controlled Trials (RCTs) tend to be non-generalizable. Little is known about the effectiveness of NPWT among typical patients. Patient registries are also ideal for assessing long term safety issues in these devices.

DETAILED DESCRIPTION:
The purpose of the Negative Pressure Wound Therapy Registry (NPWTR)) for Wounds and Ulcers is to provide comparative effectiveness data on NPWT including different NPWT devices, and safety data on NPWT (e.g. the frequency of adverse events experienced by typical NPWT patients).

NPWT promotes wound healing by applying a vacuum through a special sealed dressing. The mechanical micro-deformation of the wound bed in response to suction has been shown to stimulate and accelerate the formation of new blood vessels (angiogenesis). The continuous vacuum removes fluid and reduces edema, thereby increasing tissue oxygen levels. The vacuum may be applied continuously or intermittently, depending on the type of wound being treated and the clinical objectives. Depending on the NPWT device, a variety of dressings are placed into the wound bed in conjunction with NPWT, and a variety of suction pressures may be applied.

The diversity of NPWT devices and the rate at which they are becoming available for clinical use make it impossible to perform randomized controlled trials to compare their effectiveness against one another. Effectiveness in real world patients is the best current option to understand the role of NPWT in wound healing.

Hospital based outpatient wound centers participating in the US Wound Registry agree to provide data as part of quality initiatives including participation in PQRS, and to meet their Stage 2 Meaningful use criteria. The NPWTR is a subset of the USWR (Chronic Disease Registry) data. All patient data from all participating outpatient clinics are transmitted to the USWR where data are available for benchmarking, PQRS and other initiatives. Data used for comparative effectiveness research is HIPAA de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Provision of NPWT

Exclusion Criteria:

* patients not undergoing NPWT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing treatment with NPWT
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Healing | In days from the start of NPWT until the date healing or closure by other means, or of death from any cause, whichever came first, assessed up to 12 months
  Time-to-event for wound closure

SECONDARY OUTCOMES:
Duration of NPWT | In days from date of NPWT initiation until the date of last NPWT treatment regardless of patient outcome, assessed up to 12 months
  Counting total amount of therapy delivered
Side effects and adverse Events During Therapy | Events occurring between initial treatment and cessation of NPWT treatment. Event outcome information will be as recorded or status at 30 days following onset
  Overall catalog of event types and occurrences. Score in % for: bleeding, retention of foam or other interface in wound bed, periwound breakdown, worsening of wound such as exposure of deep structure, and wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Fife, MD, Principal Investigator — US Wound Registry
Locations (1):
- St. Luke's Wound Care Clinic, The Woodlands, Texas, United States

REFERENCES:
- [Background] Fife CE, Walker D, Thomson B, Otto G. The safety of negative pressure wound therapy using vacuum-assisted closure in diabetic foot ulcers treated in the outpatient setting. Int Wound J. 2008 Jun;5 Suppl 2(Suppl 2):17-22. doi: 10.1111/j.1742-481X.2008.00467.x. PMID 18577134
- [Background] Fife CE, Carter MJ. Wound Care Outcomes and Associated Cost Among Patients Treated in US Outpatient Wound Centers: Data From the US Wound Registry. Wounds. 2012 Jan;24(1):10-7. PMID 25875947
- [Background] Fife CE, Otto G, Walker D, Turner T, Smith L. Healing dehisced surgical wounds with negative pressure wound therapy. Ostomy Wound Manage. 2004 Apr;50(4A Suppl):28-31. No abstract available. PMID 15317243